CLINICAL TRIAL: NCT06110806
Title: Family-Based Interoceptive Exposure for Avoidant Restrictive Food Intake Disorder
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor review of inclusion/exclusion criteria and withdrawal procedures
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Robyn Sysko, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-23-00440
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Avoidant Restrictive Food Intake Disorder
Keywords: Avoidant Restrictive Food Intake Disorder; Eating Disorder; Eating Disorder Treatment; Family-Based Therapy; Exposure Therapy; Mindfulness
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: This single-site clinical trial includes non-randomizing, dose-optimizing (20 sessions) clinical trial design to examine feasibility and appropriate duration of treatment. A final assessment will take place 3-months post intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mindfulness-based interoceptive exposure (MBIE) (Experimental): Outpatient therapy for individuals with ARFID using mindfulness and exposures in a family-based therapy approach.
  Interventions: Behavioral: MBIE

INTERVENTIONS:
Behavioral: MBIE — MBIE administered over 20 sessions, targets increasing psychological flexibility and acceptance by decreasing avoidance and attempts to control distressing or undesired internal experiences, and includes psychoeducation, targeted mindfulness practice, in vivo exposures, and counter-conditioning.

SUMMARY:
This project aims to establish the feasibility and acceptability of a comprehensive mind and body intervention; specifically a mindfulness-based interoceptive exposure (MBIE) for families of youth diagnosed with avoidant/restrictive food intake disorder (ARFID). This project will: (1) explore the feasibility of recruitment, retention, and data collection procedures with youth with ARFID at end of treatment, (2) establish the acceptability and adherence of the MBIE intervention, and (3) evaluate the number of MBIE sessions required to observe changes in the number of foods avoided and mindfulness skills.

DETAILED DESCRIPTION:
A total of 57 individuals with ARFID ages 12-18 will be enrolled to outpatient mindfulness-based interoceptive exposure (MBIE). MBIE targets increasing psychological flexibility and acceptance by decreasing avoidance and attempts to control distressing or undesired internal experiences, and includes psychoeducation, targeted mindfulness practice, in vivo exposures, and counter-conditioning. MBIE will be administered in 20 sessions. Interview, self-report, anthropometrics, laboratory feeding, and behavioral task data will be used to characterize the sample to their response to treatment over time. Follow-up assessments will be completed at session 5, 10, 15, and 20. The final assessment will take place 3 months after treatment ends. Total participation will last 9 months.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* Aged 12-18
* Speaks English
* Permission from pediatrician or equivalent to receive outpatient care, including that the patient does not meet criteria for hospitalization based on the American Psychiatric Association guidelines
* Diagnosis of Avoidant Restrictive Food Intake Disorder, as assessed by the EDA-5

Parent:

* Has a child aged 12-18 with a diagnosis of ARFID
* Speaks English

Exclusion Criteria:

* Comorbid psychotic or bipolar disorder
* Psychiatric medication initiated or with a dosage change in the two weeks prior to baseline testing
* Active suicidal ideation
* Major medical condition (e.g., diabetes mellitus, pregnancy)
* Current substance dependence, as evidenced by tolerance and withdrawal
* Evidence of anatomical findings by imaging (e.g., swallow study) that would prevent safe consumption of the shake or those with a percutaneous endoscopic gastrostomy or other similar feeding tube insertion
* Children with visual or physical limitations that would preclude watching a screen and using a finger to respond with mouse clicks (e.g., blindness, epilepsy if exposure to flashing lights at certain intensities or to certain visual patterns can trigger seizures).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
MBIE-adapted Therapy Suitability and Acceptability Scale to measure Patient MBIE Therapy Tolerability | up to 6 months
  An MBIE-adapted Therapy Suitability and Acceptability Scale will average specific items from patient's view on match of therapy to the problem, responsiveness of intervention to different treatment challenges, degree of unexpected discomfort related to treatment, interest in using therapy experiences beyond the therapy session. This scale includes 10-20 items, depending on the session content, and is measured using a Likert scale from 1-7. Scores are calculated using a sum of all items, with a possible range of scores of 10 to 140. Higher scores indicate greater suitability of the treatment for the child and expectancy of success with the intervention.

SECONDARY OUTCOMES:
Therapist Adherence to MBIE Therapy | up to 6 months
  Adherence of the MBIE intervention will be measured with ratings of therapy tapes of 20 sessions. Adherence will be calculated using a dichotomous scale (yes/no) of items rating the extent of use of treatment elements and the quality of delivery of the intervention. As the number of treatment elements vary, and some items are reverse coded, the minimum, maximum, and scaling are not utilized. Per item adherence can range from 0 to 100%.
Dropout Rate | end of treatment, at approximately 6 months
  Retention will be measured using rates of dropout between baseline and session 20 (end of treatment, at approximately 6 months).
Participant Rating of Acceptability Scale | up to 9 months
  Acceptability of data collection and assessment procedures will be measured using participant ratings of acceptability for total time and frequency on an investigator-derived scale. This measurement includes items assessing the (1) tolerability and (2) ease of completing laboratory, behavior, and self-report tasks using a 15 mm visual analog scale. Scores are calculated by summing all ratings (in mm), ranging from 0-20. Higher scores indicate greater acceptability of study assessments.
Functional Food Hierarchy to Measure Tolerability | up to 6 months
  The number of MBIE sessions required to achieve a clinically meaningful outcome and acceptable tolerability using a Functional Food Hierarchy. This measurement rates a minimum of 11 food items on a scale of 0-10 at 10 levels of the hierarchy (subjective units of distress). Scores range from 0-100 with higher scores indicating lower avoidance/increased consumption.
Number of MBIE sessions required to achieve tolerability | up to 6 months
  The number of MBIE sessions required to achieve a clinically meaningful outcome (consuming food rated as70 or higher on the Food Avoidance Scale). The Food Avoidance Scale is investigator-derived and includes 1 item rated on a scale of 0-100 with higher scores indicating consumption of more challenging/avoided foods.
Change in total calories consumed | Baseline and approximately 10 weeks
  Autonomous eating will be measured in total calories consumed during a single-item meal. Total calories consumed will be calculated between baseline and session 10 of treatment
Change in total calories consumed | Baseline and approximately 6 months
  Autonomous eating will be measured in total calories consumed during a single-item meal. Total calories consumed will be calculated between baseline and end of treatment (session 20).
Change in Expected Body Weight Percentage | Baseline and approximately 6 months
  Expected body weight percentage will be calculated for age and sex to evaluate physical status at baseline and end of treatment (session 20) to evaluate any changes during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Sysko, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Department of Psychiatry, Eating and Weight Disorders Program, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Twice yearly
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  Any purpose. Specify Other Mechanism Data will be made available through the National Institute of Mental Health Data Archive (NDA)